CLINICAL TRIAL: NCT00179010
Title: Use of AMP to Improve Tissue Delivery of Adenosine
Brief Title: AMP as a Better Delivery System of Adenosine
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study was terminated because funding could not be secured
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Italo Biaggioni, Professor of Medicine, Vanderbilt University Medical Center
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 030371
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Results first posted 2019-05-07 (Actual); Last update posted 2019-05-07 (Actual); Status verified 2019-05

CONDITIONS: Ischemia
Keywords: Adenosine; AMP; Microdialysis; Blood Flow
MeSH Terms: conditions — Ischemia | interventions — Adenosine; beta-apocarotenoid-14',13'-dioxygenase; Adenosine Monophosphate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Adenosine then Adenosine Mono Phosphate (AMP) (Experimental): Intrarterial infusion of adenosine then same subject switch to AMP one month apart.
  Interventions: Drug: Adenosine; Drug: Adenosine Mono Phosphate (AMP)
- Adenosine Mono Phosphate (AMP) then adenosine (Experimental): Intrarterial infusion of AMP then same subject switch to Adenosine one month apart.
  Interventions: Drug: Adenosine; Drug: Adenosine Mono Phosphate (AMP)

INTERVENTIONS:
Drug: Adenosine — Adenosine intrarterial (intrabrachial) infusion at 3 diferent doses for 15 minutes each
  Other Names: Ado
Drug: Adenosine Mono Phosphate (AMP) — Intraterial infusion of AMP at 3 different doses for 15 minutes each (at equimolar doses as adenosine)
  Other Names: AMP

SUMMARY:
Adenosine and AMP are substances normally present in the body. Adenosine is also given for the treatment of some heart rhythm problems and may be used to reduce heart damage during heart attacks. The problem in using adenosine is that it is taken up by cells and, therefore, very little of the adenosine we give by vein or in the artery actually reaches the tissue. We propose to use AMP as a way to improve delivery of adenosine. AMP is inactive by itself, but is converted to adenosine in tissue. We hope that by giving AMP we will increase levels of adenosine in tissue. To see if this is true, we will give either adenosine or AMP into the forearm artery while we measure how much adenosine reaches the forearm tissue.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* Age 18-65
* Non smokers

Exclusion Criteria:

* Smokers
* Any chronic disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2003-10; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Italo Biaggioni, M.D., Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited through mass e-mails and flyers posted in campus
Pre-assignment Details: Subjects were randomly assigned to each treatment arm, after being screened for any medical problem that would be considered a contraindication for the study according to the physician performing the initial evaluation. Once subjects completed one arm, they were crossed to the other arm and studied at lest one month after.
Groups:
- Adenosine First Then AMP: Intrarterial infusion of adenosine first
  Adenosine: Adenosine intrarterial (intrabrachial) infusion at 3 diferent doses for 15 minutes each
  Subjects in this group were assigned to received intrarterial infusions of adenosine and then crossed to the other arm (AMP) after at least 1 month.
- Adenosine Mono Phosphate (AMP) First Then Adenosine: Intrarterial infusion of AMP first
  Adenosine Mono Phosphate (AMP): Intraterial infusion of AMP at 3 different doses for 15 minutes each (at equimolar doses as adenosine)
  Subjects intros group were assigned to received intrarterial infusions of AMP and then crossed to the other arm (adenosine), at least 1 month after.
Period: Overall Study
Arm/Group | Adenosine First Then AMP | Adenosine Mono Phosphate (AMP) First Then Adenosine
Started | 6 | 7
Completed | 5 | 5
Not Completed | 1 | 2
Not completed — Muscle probe defective | 1 | 1
Not completed — Failure to place arterial line | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Adenosine Mono Phosphate (AMP) First: Intrarterial infusion of AMP
  Adenosine Mono Phosphate (AMP): Intraterial infusion of AMP at 3 different doses for 15 minutes each (at equimolar doses as adenosine)
- Adenosine First: Intrarterial infusion of adenosine
  Adenosine: Adenosine intrarterial (intrabrachial) infusion at 3 diferent doses for 15 minutes each
- Total: Total of all reporting groups
Arm/Group | Adenosine Mono Phosphate (AMP) First | Adenosine First | Total
Number analyzed (Participants) | 7 | 6 | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 6 | 13
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 37 (10) | 37 (10) | 37 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 4 | 3 | 7
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7 | 6 | 13

OUTCOME MEASURES:

1. Primary Outcome: Interstitial Adenosine Levels
Time Frame: Microdyalysis samples for adenosine, were collected for 15 minutes at each stage of the study (baseline and each dose of adenosine or AMP)
Population: 13 subjects received both treatments. 3 subject did not complete the study and were excluded. We are reporting data in only 10 subjects that have collected samples.
Measure: Mean (Standard Error); unit: nM
Groups:
- Adenosine: Intrarterial infusion of adenosine
  Adenosine: Adenosine intrarterial (intrabrachial) infusion at 3 diferent doses for 15 minutes each
- Adenosine Mono Phosphate (AMP): Intra-arterial infusion of AMP
Arm/Group | Adenosine | Adenosine Mono Phosphate (AMP)
Number analyzed (Participants) | 10 | 10
nM
  Third dose | 93.2 (15.7) | 91.7 (13.8)
  Second Dose | 87.5 (12.7) | 91.1 (18.9)
  First Dose | 89.8 (18.6) | 86.2 (13.9)
Statistical Analysis 1: Comparison: Adenosine; Test type: Superiority or Other; p = 0.854, ANOVA

2. Other Pre Specified Outcome: Forearm Blood Flow
Time Frame: End of each stage (minute 15) of the study (baseline and each dose of adenosine or AMP ia infusions)
Population: This was an exploratory Outcome and was abandoned.
Groups:
- Adenosine Mono Phosphate (AMP): Intrarterial infusion of AMP
  Adenosine Mono Phosphate (AMP): Intraterial infusion of AMP at 3 different doses for 15 minutes each (at equimolar doses as adenosine)
Arm/Group | Adenosine | Adenosine Mono Phosphate (AMP)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Adenosine | Adenosine Mono Phosphate (AMP)
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 0/13 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No